CLINICAL TRIAL: NCT06465147
Title: REACT-01: Reversing Autoimmunity Through Cell Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director & Co-Chief Medical Officer, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REACT-01
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: CAR T cells; Lupus; Systemic Lupus Erythematosus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SCRI-CAR19v3 (Experimental): Single infusion of SCRI-CAR19v3
  Interventions: Biological: SCRI-CAR19v3

INTERVENTIONS:
Biological: SCRI-CAR19v3 — Single infusion of SCRI-CAR19v3

SUMMARY:
This is a phase 1, open-label, non-randomized study enrolling pediatric and young adult research participants with treatment-refractory Systemic Lupus Erythematosus (SLE), to examine the safety, feasibility, and efficacy of administering T cell products derived from peripheral blood mononuclear cells (PBMC) that have been genetically modified to express CD19 specific chimeric antigen receptor (CAR)

A child or young adult meeting all eligibility criteria and meeting none of the exclusion criteria will have their T cells collected. The T cells will then be bioengineered into a CAR T cell that targets circulating and tissue residing B cells.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 2-30 years old. The first 3 subjects will be aged ≥ 17. The FDA will review safety data to determine if the age can be lowered first to ≥ 12 then, following the treatment of 3 further subjects aged 12-17, to ≥ 2
* Serologically active Systemic Lupus Erythematosus that is refractory to treatment
* Able to tolerate apheresis or already has an apheresis product available for use in manufacturing.
* ≥ 24 weeks post last Rituximab or related B cell depleting therapy
* ≥ 12 weeks post last Belimumab / Anifrolumab therapy
* ≥ 4 weeks post last calcineurin inhibitor treatment
* For subjects receiving non-calcineurin immunosuppressive therapy, on a stable dose for ≥ 8 weeks before enrollment
* For subjects receiving corticosteroid therapy, on a stable dose for ≥ 2 weeks before enrollment
* Adequate organ function
* Adequate laboratory values
* Subjects of childbearing or child-fathering potential must agree to use highly effective contraception from consent through 12 months following infusion of investigational product on trial
* Subjects must be willing to remain within 1 hour's drive of Seattle Children's Hospital for 4 weeks following CAR T cell infusion.
* Subject and/or legally authorized representative has signed the informed consent form for this study

Exclusion Criteria:

* History or presence of active CNS lupus or other CNS disease
* Kidney dysfunction requiring renal replacement therapy
* Pregnant or breastfeeding
* Insufficient pulmonary reserve including history of COPD, >10 pack year smoking history or SLE lung disease with hypoxia at rest with oxygen saturation ≤92% on room air
* Unable to tolerate repletion with any formulation of IgG.
* Active or prior malignancy, unless the malignancy was treated and there is no evidence of recurrent disease <5 years from enrollment.
* Prior solid organ transplantation.
* Presence of an active severe infection
* Presence of any condition that, in the opinion of the investigator, would prohibit the subject from undergoing treatment under this protocol

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2041-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 days post-infusion
  The investigators will assess and described the type, frequency, severity, and duration of adverse events associated with the CAR T cell product.
Rate of SCRI-CAR19v3 Manufacturing Success | 28 days
  We will measure the number of successfully manufactured SCRI-CAR19v3 products.

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Jackson, MD, Study Chair — Seattle Children's Hospital; Colleen Annesley, MD, Study Director — Seattle Children's Hospital; Corinne Summers, MD, Study Director — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States